CLINICAL TRIAL: NCT00252954
Title: Effects of Levetiracetam on Chronic Neuropathic Pain Following Spinal Cord Injury: a Randomized, Double-blind, Placebo-controlled, Cross-over, Multi-center Study
Brief Title: Levetiracetam in Chronic Neuropathic Pain Following Spinal Cord Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Collaborators: UCB Nordic A/S (Industry)
Responsible Party: Nanna Brix Finnerup, Danish Pain Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LEV-2005
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Injuries, Spinal Cord; Pain
Keywords: Spinal cord injury; Neuropathic pain; Spasms
MeSH Terms: conditions — Spinal Cord Injuries; Pain; Neuralgia; Spasm | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Placebo Comparator)
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Tablets 2000-3000 mg per day

SUMMARY:
Purpose: To evaluate the efficacy and safety of levetiracetam on chronic neuropathic pain after spinal cord injury, and to examine its effect on spasms and evoked pain.

DETAILED DESCRIPTION:
Study design: Randomized double-blind cross-over study of levetiracetam (Keppra) against corresponding placebo with a 1 week baseline period followed by 2 x 5 weeks treatment periods separated by a 1 week wash-out period.

Methodology: Levetiracetam and corresponding placebo is gradually increased during two weeks from 500 mg x 2 daily to 1500 mg x 2 daily (1000 mg x 2 daily is allowed if 1500 mg x 2 is not tolerated), and kept on that dose for three weeks.

The study will be monitored by the GCP units of Aarhus and Copenhagen University.

ELIGIBILITY:
Inclusion Criteria:

* 1. age 18 or more
* 2. neuropathic pain (that have lasted at least 3 month) after a spinal cord injury with a pain intensity of at least 4 on a 0-10 point numeric rating scale

Exclusion Criteria:

* 1. pregnancy or lactation
* 2. allergy to levetiracetam
* 3. alcohol or substance abuse, mental disease, epilepsy, depression and psychiatric disorders, severe liver disease, decreased kidney function, and known concomitant cerebral damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-11; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in median pain intensity (measured daily on a 10 point NRS) of spontaneous pain from baseline week to last week of treatment. | Last week of each 5-week treatment period

SECONDARY OUTCOMES:
Spasms and spasticity; pain relief for total, at- and below-level pain; evoked pain; escape medication; NPSI; predictive value of the presence of evoked pain; Global impression of change; sleep disturbance. | Last day of each 5-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Nanna B Finnerup, MD, Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Danish Pain Research Center, Aarhus University Hospital, Aarhus
  - Clinic for Spinal Cord Injuries, Rigshospitalet, Hornbæk
  - The Spinal Cord Unit, Dept of Rheumatology, Viborg

REFERENCES:
- [Derived] Finnerup NB, Grydehoj J, Bing J, Johannesen IL, Biering-Sorensen F, Sindrup SH, Jensen TS. Levetiracetam in spinal cord injury pain: a randomized controlled trial. Spinal Cord. 2009 Dec;47(12):861-7. doi: 10.1038/sc.2009.55. Epub 2009 Jun 9. PMID 19506571